CLINICAL TRIAL: NCT07191587
Title: Vitamin B Prophylaxis Effect on Peripheral Neuropathy Induced in Ovarian Cancer Patients Receiving Paclitaxel Based Regimen.
Brief Title: A Controlled Clinical Trial Assessing the Efficacy of Vitamin B Prophylaxis in Attenuating Paclitaxel-induced Neuropathy and the Imperative Use of Gabapentin in Diabetic Ovarian Cancer Patients and the Potential Effect on Disease Response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MO2411-505-068-193
Record Dates: First submitted 2025-09-02; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Neuropathy, Chemotherapy-induced; Disease Management
Keywords: Vitamin B; Paclitaxel-induced peripheral neuropathy; Ovarian cancer; Diabetic; Gabapentin
MeSH Terms: conditions — Peripheral Nervous System Diseases; Ovarian Neoplasms | interventions — Vitamin B Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic arm (Active Comparator): In this arm, patients were given oral vitamin B prophylaxis prior to their first cycle of chemotherapy.
  Interventions: Dietary Supplement: Vitamin B Complex
- Non-prophylactic arm (Other): In this arm, patients were given oral vitamin B upon developing chemotherapy-induced peripheral neuropathy.
  Interventions: Dietary Supplement: Vitamin B Complex

INTERVENTIONS:
Dietary Supplement: Vitamin B Complex — Vitamin B complex given as prophylaxis in prophylactic arm and as treatment in non-prophylactic arm.

SUMMARY:
The goal of this clinical trial is to learn if vitamin B prophylaxis is effective in attenuating chemotherapy-induced peripheral neuropathy in adult ovarian cancer patients. The main questions (primary outcomes) it aims to answer are:

* The severity of chemotherapy-induced peripheral neuropathy in ovarian cancer patients undergoing a weekly paclitaxel-based regimen in the vitamin B prophylactic group versus non-prophylactic group.
* Severity of chemotherapy-induced peripheral neuropathy in diabetic patients versus non-diabetic patients in both prophylactic and non-prophylactic groups.

Participants will:

Take drug oral vitamin B complex every day as prophylaxis for 6 months. Visit the clinic once every week for their weekly Paclitaxel regimen, checkups and tests.

Keep a diary of their symptoms.

DETAILED DESCRIPTION:
Patients received oral vitamin B complex as prophylaxis prior to starting their paclitaxel-based regimen and patients in the non-prophylaxis group received oral vitamin B complex upon developing chemotherapy-induced peripheral neuropathy during their treatment with paclitaxel-base regimen. Gabapentin was given to the patients in either groups upon aggravation of CIPN symptoms whether in severity or neuropathic pain according to peripheral neuropathy grading.

Secondary outcomes:

* The number of patients in both prophylactic and non-prophylactic groups who required Gabapentin upon uncontrolled or aggravation in CIPN with vitamin B complex only.
* Impact of vitamin B complex prophylaxis on dose modification of paclitaxel-based regimen.
* Association between dose modification and CA 125 status.
* Progression-free survival (PFS) was evaluated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with confirmed pathology of ovarian adenocarcinoma.
* Aged 18 years or older.
* Scheduled to receive a weekly paclitaxel-based chemotherapy regimen (80 mg/m²).

Exclusion Criteria:

* Individuals under 18 years of age.
* Any patients with pre-existing peripheral neuropathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Severity of chemotherapy-induced peripheral neuropathy (peripheral neuropathy grade) | At baseline and up to 18 weeks.
  The primary outcome of this study was the severity of chemotherapy-induced peripheral neuropathy in ovarian cancer patients undergoing a weekly paclitaxel-based regimen in the vitamin B prophylactic group versus non-prophylactic group. Severity was assessed by assessed by CTCAE v4.0 through monitoring the occurrence of peripheral neuropathy symptoms (peripheral neuropathy grade) at baseline and on weekly basis, up to 18 weeks (last follow up for chemotherapy induced peripheral neuropathy).

SECONDARY OUTCOMES:
Number of participants with paclitaxel induced peripheral neuropathy as assessed by CTCAE v4.0 in both prophylactic and non-prophylactic groups who required Gabapentin upon uncontrolled or aggravation in neuropathy grade with vitamin B complex only. | After the first week and up to 18 weeks.
Severity of chemotherapy-induced peripheral neuropathy (peripheral neuropathy grade) as assessed by CTCAE v4.0 in diabetic patients versus non-diabetic patients in both prophylactic and non-prophylactic groups. | At baseline and up to 18 weeks.
Percentage of patients that underwent dose modification in their paclitaxel regimen in both prophylactic and non-prophylactic groups due to chemotherapy-induced peripheral neuropathy as assessed by CTCAE v4.0". | After the first week and up to 18 weeks.
Association between dose modification in paclitaxel regimen and CA125 status as measured by improved or worsened CA125 status. | up to 20 weeks.
  The CA125 status after dose modification in paclitaxel regimen due to chemotherapy-induced peripheral neuropathy or other hematological toxicities.
Progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Diabetes mellitus as a risk factor for chemotherapy-induced peripheral neuropathy: a meta-analysis — https://doi.org/10.1007/s00520-021-06321-7
- See also: Vitamin B6 status and chronic chemotherapy-induced peripheral neuropathy: a prospective cohort study among patients with non-metastatic colorectal cancer receiving oxaliplatin-based chemotherapy — https://doi.org/10.1136/bmjonc-2024-000462